CLINICAL TRIAL: NCT02642783
Title: Sensory Evaluation of Laxative Bowel Solutions Used Prior to Colonoscopy
Brief Title: Sensory Properties of Bowel Cleansing Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ammar Olabi, Associate Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NUT.AO.19
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Laxative Bowel Cleansing Solutions
Keywords: laxatives; sensory evaluation; acceptability; colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Descriptive analysis (Other): panelists were asked to rate different sensory attributes for different laxative bowel cleansing solutions on a 15 cm line scale.
  Interventions: Behavioral: Descriptive analysis
- Acceptability test (Other): panelists were asked to rate the acceptability of different laxative bowel cleansing solutions using the 9-point hedonic scale.
  Interventions: Behavioral: acceptability test

INTERVENTIONS:
Behavioral: Descriptive analysis — subjects were asked to assess the sensory profile by tasting the laxative bowel cleansing solutions, namely: Moviprep, picoprep, fortrans and isinova
  Arms: Descriptive analysis
Behavioral: acceptability test — subjects were asked to assess the acceptability of the laxative bowel cleansing solutions, namely: Moviprep, picoprep, fortrans and isinova
  Arms: Acceptability test

SUMMARY:
Samples of 4 commercially available bowel cleansing solutions, namely PEG-electrolyte + ascorbic acid (PEG-Asc, Moviprep®, Norgine, UK), PEG-electrolyte (PEG, Fortrans® Ibsen, France), sodium picosulfate/magnesium citrate (SPS, Picoprep®, Ferring, Switzerland), and oral sodium sulfate (OSS, Izinova®, Ibsen, France) were prepared according to the manufacturer's instructions. Descriptive analysis was conducted with trained panelists (N= 14) to create a sensory profile for the solutions and generated attributes were rated on an unstructured 15-cm line scale using the Compusense at-hand® (Guelph, Canada) sensory evaluation software. Acceptability testing was carried out with untrained participants (N=80) and samples were rated on the 9-point hedonic scale. Moreover, a Just-About-Right (JAR) scale was included for the four basic tastes to determine their compatibility with optimum taste/acceptability levels in the products.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years

Exclusion Criteria:

* allergies to polyethelene glycol (PEG), artificial sweeteners

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
rating of sensory attributes | 3 weeks
  participants attended 4 training sessions during which they generated sensory descriptive attributes specific for the tasted laxative solutions. In addition, they evaluated the laxative samples by rating generated attributes on a 15-cm unstructured line scale using compusense at-hand sensory evaluation software.

SECONDARY OUTCOMES:
Acceptability Score | 1 week
  untrained participants evaluated the laxative samples for acceptability testing using the 9-point hedonic scale.
Just about right score | 1 week
  Participants evaluated the laxative samples for the 4 basic tastes (saltiness, sourness, sweetness and bitterness) to determine their compatibility with optimum taste levels in the products.

IPD SHARING:
Plan to Share IPD: No